CLINICAL TRIAL: NCT03859869
Title: Creon (Pancrelipase) Therapy for Subjects With Exocrine Pancreatic Insufficiency (EPI) Due to Pancreatic Cancer: A Double-blind, Randomized, Parallel Design With 2 Dose Cohorts of Pancrelipase in Resected Pancreatic Cancer Subjects and an Open-label Single Dose Cohort in Non-resected Pancreatic Cancer Subjects
Brief Title: A Study of Creon (Pancrelipase) in Resected and Non-resected Pancreatic Cancer Participants With Exocrine Pancreatic Insufficiency (EPI)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Considerations (difficulty with enrollment)
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-142
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Exocrine Pancreatic Insufficiency (EPI)
Keywords: Exocrine Pancreatic Insufficiency (EPI); Pancreatic Cancer; Creon; Pancrelipase
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Pancreatic Neoplasms | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Resected Participants Receiving Low Dose (12,000/6,000 units lipase) Pancrelipase (Experimental): Resected participants (surgery to remove pancreatic cancer) will first be given low dose pancrelipase. Low dose is defined as 12,000 USP units (lipase) with meals and 6000 U with snacks. At Weeks 1, 5, or 9, participants will be evaluated, and those who meet criteria for dose increase will be given high dose pancrelipase. High dose is defined as 72,000 U with meals and 36,000 U with snacks. All participants will receive placebo as needed to keep the number of pills the same in each group and for blinding.
  Interventions: Drug: Pancrelipase; Drug: Placebo
- Resected Participants Receiving High Dose (72,000/36,000 units lipase) Pancrelipase (Experimental): Resected participants (surgery to remove pancreatic cancer) will receive and continue on high dose pancrelipase throughout the study. High dose is defined as 72,000 USP units (lipase) with meals and 36,000 U with snacks. All participants will receive placebo as needed to keep the number of pills the same in each group and for blinding.
  Interventions: Drug: Pancrelipase; Drug: Placebo
- Non-Resected Participants Receiving High Dose (72,000/36,000 units lipase) Pancrelipase (Experimental): Non-resected participants (those who did not have surgery to remove pancreatic cancer) will receive high dose pancrelipase throughout the study in an open-label cohort. High dose is defined as 72,000 USP units (lipase) with meals and 36,000 U with snacks.
  Interventions: Drug: Pancrelipase

INTERVENTIONS:
Drug: Pancrelipase — Pancrelipase is administered orally as capsules with a meal or snack
  Other Names: Creon
Drug: Placebo — Placebo is administered orally as capsules with a meal or snack
  Arms: Resected Participants Receiving High Dose (72,000/36,000 units lipase) Pancrelipase; Resected Participants Receiving Low Dose (12,000/6,000 units lipase) Pancrelipase

SUMMARY:
This is a study in participants with Exocrine Pancreatic Insufficiency (EPI) due to pancreatic cancer. This study will include resected participants who are post pancreatic cancer surgery, and an additional cohort in non-resected participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant has diagnosed cancer of pancreas with biopsy and/or radiography, with a life expectancy of at least 5 months at screening
* Participant's pancreatic cancer must involve the head and/or neck of the pancreas
* Confirmed exocrine pancreatic insufficiency (EPI) as evidenced by fecal elastase-1 (FE-1) ≤ 150 µg/g stool at screening
* A positive Sudan stain for participants without history of fat malabsorption (fat malabsorption is defined as clinical steatorrhea, or measured stool fat > 7 g/day, or positive stool results by Sudan stain) within 1 week of screening -- Positive stool results are defined as increased level of neutral OR total fats

Exclusion Criteria:

* Participant has neuroendocrine pancreatic cancer
* Participant has fibrosing colonopathy
* Participant has any other malignancy within 1 year of screening
* Participant has uncontrolled gout, including those with a recent flare within 60 days of screening
* Participant has other significant organ or bone marrow abnormality within 60 days of screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (33):
- United States (33):
  - Alabama Oncology /ID# 207770, Birmingham, Alabama
  - Banner University of Arizona Medical Center Phoenix /ID# 208402, Phoenix, Arizona
  - UCSF Fresno /ID# 205757, Fresno, California
  - Stanford University School of Med /ID# 208821, Stanford, California
  - UCH-MHS Memorial Hospital Central /ID# 207093, Colorado Springs, Colorado
  - UCHealth Cancer Care and Hematology Clinic /ID# 207091, Fort Collins, Colorado
  - George Washington University Medical Faculty Associates /ID# 203363, Washington D.C., District of Columbia
  - University of Florida - Archer /ID# 202679, Gainesville, Florida
  - Columbus Regional Research Institute /ID# 211394, Columbus, Georgia
  - Northwest Community Hospital /ID# 202270, Arlington Heights, Illinois
  - NorthShore University HealthSystem /ID# 209026, Evanston, Illinois
  - Ingalls Memorial Hosp /ID# 203962, Harvey, Illinois
  - Advocate Christ Medical Center /ID# 203132, Oak Lawn, Illinois
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 204407, Ann Arbor, Michigan
  - Ascension Providence Hospital /ID# 203449, Southfield, Michigan
  - St. Louis University /ID# 205769, St Louis, Missouri
  - Mercy Hospital South /ID# 221766, St Louis, Missouri
  - Northwell Health Center for Liver Diseases /ID# 207321, Manhasset, New York
  - NYU Winthrop Hospital /ID# 207513, Mineola, New York
  - New York University Langone Me /ID# 202290, New York, New York
  - Columbia University Medical Center /ID# 204165, New York, New York
  - East Carolina University /ID# 206661, Greenville, North Carolina
  - Gabrail Cancer Center Research /ID# 208030, Canton, Ohio
  - Ohio State Cancer Center /ID# 203131, Columbus, Ohio
  - Fox Chase Cancer Center /ID# 202288, Philadelphia, Pennsylvania
  - Reading Hospital /ID# 206869, Reading, Pennsylvania
  - Musc /Id# 210727, Charleston, South Carolina
  - Tennessee Cancer Specialists /ID# 208235, Knoxville, Tennessee
  - Vanderbilt University Medical Center /ID# 204231, Nashville, Tennessee
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 206156, Dallas, Texas
  - UT MD Anderson Cancer Center /ID# 202271, Houston, Texas
  - Wisconsin Center for Advanced Research, a division of GI Associates, LLC /ID# 205746, Milwaukee, Wisconsin
  - Medical College of Wisconsin /ID# 205714, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link: https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Neither the Resected Participants Receiving Low Dose Pancrelipase group nor the Non-Resected Participants Receiving High Dose Pancrelipase group enrolled any participants.
Period: Overall Study
Arm/Group | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase | Non-Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase
Started | 0 | 1 | 0
Completed | 0 | 1 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase | Non-Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase | Total
Number analyzed (Participants) | 0 | 1 | 0 | 1
Age, Customized [Count of Participants; unit: Participants]
  Age 21 - 90 years old | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 0 |  | 0
  Male |  | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  | 0
  Asian |  | 0 |  | 0
  Native Hawaiian or Other Pacific Islander |  | 0 |  | 0
  Black or African American |  | 0 |  | 0
  White |  | 1 |  | 1
  More than one race |  | 0 |  | 0
  Unknown or Not Reported |  | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Stool Fat From Baseline (Day 1) to Week 1 (Day 8) Among Participants With Resected Pancreatic Cancer
Description: Stool samples were collected during the 48 hours prior to the Day 1 and Week 1 visits and analyzed for fat content.
Time Frame: Baseline (Day 1), Week 1 (Day 8)
Population: Participants who received at least one dose of study drug and who had evaluable stool fat at both Baseline and Week 1 visits
Measure: Mean (Standard Deviation); unit: g/24 hours
Arm/Group | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase
Number analyzed (Participants) | 0 | 1
g/24 hours |  | 3.1

2. Secondary Outcome: Change in Average Daily Stool Frequency From Baseline (Day 1) to Week 1 (Day 8) Among Participants With Resected Pancreatic Cancer
Description: Participants recorded stool frequency using an electronic diary (eDiary). The average daily stool frequency was calculated from the last 3 days prior to the Baseline and Week 1 visits.
Time Frame: Baseline (Day 1), Week 1 (Day 8)
Population: Participants who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: number of stools/day
Arm/Group | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase
Number analyzed (Participants) | 0 | 1
number of stools/day |  | NA — Not calculable/estimable because stool frequency data for Week 1 is missing

3. Secondary Outcome: Change in Stool Consistency From Baseline to Week 1 Among Participants With Resected Pancreatic Cancer
Description: Participants recorded stool consistency using an electronic diary (eDiary). The change from Baseline to Week 1 is the proportion of days having watery stool consistency in the last 7 days prior to each of Baseline and Week 1 visits. Negative changes from Baseline indicate less frequent watery stools.
Time Frame: Baseline (Day 1), Week 1 (Day 8)
Population: Participants who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: proportion of days w/ watery consistency
Arm/Group | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase
Number analyzed (Participants) | 0 | 1
proportion of days w/ watery consistency |  | -0.29

4. Secondary Outcome: Change in the Total EPI Symptoms Score From Baseline to Week 1 Among Participants With Resected Pancreatic Cancer
Description: The EPI Symptoms Questionnaire consists of 12 questions. The response scores range from 0 to 4 for each question (0 corresponding to None to 4 corresponding to Very Severe), with the total score ranging from 0 to 48. Positive changes indicate worsening from Baseline.
Time Frame: Baseline (Day 1), Week 1 (Day 8)
Population: Participants who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase
Number analyzed (Participants) | 0 | 1
units on a scale |  | 3

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; time on follow up was 161 days. TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; time on study drug was 92 days.
Description: Neither the "Resected Participants Receiving Low Dose (12,000/6,000 units lipase) Pancrelipase" group nor the "Non-Resected Participants Receiving High Dose (72,000/36,000 units lipase) Pancrelipase" group enrolled any participants.
Arm/Group | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase | Non-Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resected Participants Receiving Low Dose (12,000/6,000 Units Lipase) Pancrelipase (N=0) | Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase (N=1) | Non-Resected Participants Receiving High Dose (72,000/36,000 Units Lipase) Pancrelipase (N=0)
WHITE BLOOD CELLS DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 0 (0)
POSTURAL DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated due to low enrollment rates. The decision to terminate the study was not based on any safety or efficacy data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03859869/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT03859869/SAP_001.pdf